CLINICAL TRIAL: NCT06015633
Title: Exploration of Ocular, Vascular, and Genetic Findings Associated and Correlated with the Presence of Late-stage AMD
Brief Title: Ocular, Vascular, and Genetic Findings in AMD Patients
Status: Active, not recruiting | Type: Observational
Sponsor: OcuDyne, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OC-2301TV
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Exudative AMD: Subjects that have at least one eye with a history of, or active, exudative age related macular degeneration
  Interventions: Other: No intervention
- Non-exudative AMD: Subjects that have at least one eye with late stage non-exudative age-related macular degeneration (presence of geographic atrophy)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational only

SUMMARY:
Observation of findings associated with AMD

DETAILED DESCRIPTION:
Explorational observation of ocular, vascular, and genetic findings in patients diagnosed with AMD

ELIGIBILITY:
Inclusion Criteria:

1. At least 55 years of age at the time of consent
2. Able to understand and provide written informed consent
3. Sufficiently clear ocular media, adequate pupillary dilation, and adequate fixation to permit quality fundus imaging
4. Able to cooperate with ophthalmic visual function testing and anatomic assessments
5. Diagnosed with late-stage AMD in at least one eye. (if both eyes of an eligible subject meet inclusion criterion, the more advanced eye will receive primary eye assignment)
6. Willing to have protocol specified genetic testing
7. Willing to have head coil MRI/A (with contrast if deemed necessary)

Exclusion Criteria:

Ocular

1. History of any retinal disease other than AMD in either eye
2. Spherical equivalent refractive error demonstrating >6 diopters of myopia or an axial length >26 mm in the study eye
3. History of vitrectomy in the study eye
4. Any intraocular surgery (including lens replacement surgery) in the study eye, within 90 days of enrollment
5. History of endophthalmitis
6. Trabeculectomy or aqueous shunt or valve in the study eye
7. Aphakia or absence of the posterior capsule in the study eye (Note: Previous violation of the posterior capsule is also excluded unless it occurred as a result of yttrium aluminum garnet [YAG] laser posterior capsulotomy in association with prior posterior chamber intraocular lens implantation and at least 90 days prior to enrollment)
8. Presence of advanced guttae or visually significant keratopathy that would cause scattering of light or alter visual function in the study eye
9. History of idiopathic or autoimmune-associated uveitis in either eye
10. Active inflammation or infection, including conjunctivitis, keratitis, or scleritis in either eye
11. GA secondary to a condition other than AMD (e.g., Stargardt's disease, cone rod dystrophy, or toxic maculopathies such as Plaquenil maculopathy) in either eye

    Non-Ocular
12. Use of any investigational product or investigational medical device (i.e., not approved by FDA for the specific use) within 90 days prior to screening or anticipated use during the study
13. Women of childbearing potential who are pregnant or unwilling to use effective contraception for the duration of the study
14. Acute or serious illness, in the opinion of the site investigator
15. History of kidney failure or gadolinium toxicity

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with exudative or non-exudative late-stage age-related macular degeneration.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
OCT-A | Baseline observation of incidence / correlation only
  OCT-A metrics in subjects with AMD

SECONDARY OUTCOMES:
Genetic markers related to AMD | Baseline observation of incidence / correlation only
  Presence of 52 known AMD related genetic markers
Magnetic Resonance Angiography | Baseline observation of incidence / correlation only
  Ophthalmic artery MRI / MRA results in subjects with AMD

CONTACTS AND LOCATIONS:
Overall Officials: Luana Wilbur, BS, Study Director — OcuDyne VP, Clinical and Regulatory Affairs
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No